CLINICAL TRIAL: NCT04480775
Title: Triamcinolone Versus Methylprednisolone in Ultrasound Guided Transversus Abdominis Plane Block in Major Open Abdominal Surgery
Brief Title: Triamcinolone Versus Methylprednisolone in Transversus Abdominis Plane Block
Acronym: triamcinolone
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: ghada fouad (Other)
Responsible Party: Sponsor-Investigator, ghada fouad, associate professor, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: (MS.20.01.999-2020/01/10)
Record Dates: First submitted 2020-07-13; First posted 2020-07-21 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Major Abdominal Surgery
Keywords: triamicinolone; methylprednisolone; transversus abdominisus plane block
MeSH Terms: interventions — Triamcinolone; Methylprednisolone; Bupivacaine

STUDY DESIGN:
Intervention Model Description: Patient will be evaluated pre operative and full lab will be done In the Pre Anaesthesia Room ,a 20 gauge venous catheter will be inserted in the upper limb , and monitoring included heart rate, electrocardiogram, noninvasiveblood pressure, and peripheral oxygen saturation.Oxygen at the rate of 6 L/min will beadministered through oxygen mask to all patients.
  The anesthesiologist who performed the block will be blinded to drug solution and not involved in data collection, another anesthesiologist will prepare drug solution and other anesthesiologist collect the data.
Who Masked: Participant, Investigator
Masking Description: double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- bupivacaine group (Experimental): 28 Patients will receive 18 ml of bupivacaine 0.5 % plus 1ml 0.9% saline in TAP block divided equally on both sides
  Interventions: Drug: bupivacaine
- triamicinolone group (Active Comparator): 28 Patient will receive 18 ml of bupivacaine 0.5 % plus (20 mg of triamcinolone in 1ml 0.9% saline divided equally on both sides in TAP block
  Interventions: Drug: Triamcinolone; Drug: bupivacaine
- methylprednisolone group (Active Comparator): 28 Patient will receive 18 ml of bupivacaine 0.5 % plus (40 mg of methylprednisolone in 1ml 0.9% saline ) on both sides in TAP block.
  Interventions: Drug: Methylprednisolone; Drug: bupivacaine

INTERVENTIONS:
Drug: Triamcinolone — transversus abdominis plane block with bupivacain and triamicinolone
  Arms: triamicinolone group
Drug: Methylprednisolone — transversus abdominis plane block with bupivacaine and methylprednisolone
  Arms: methylprednisolone group
Drug: bupivacaine — transversus abdominis plane block with bupivacaine alone

SUMMARY:
In the current Study we will compare between triamcinolone and methylprednisolone as an additive to bupivacaine drug in ultrasound guided TAP block in major open abdominal surgery .

DETAILED DESCRIPTION:
Postoperative pain is one of the main causes of respiratory function derangement after abdominal surgery .Transversus abdominis plane (TAP) block is widely used in abdominal surgery for postoperative analgesia The transversus abdominis plane (TAP) block is aperipheral nerve block that involves the injection of alocal anesthetic (LA) in the plane between the internaloblique and transversus abdominis muscle layers, with the aim of anesthetizing the intercostal nerves supplyingthe abdominal wall (from T6 to L1) By blocking intercostal nerves T6 to L1, TAPblock efficiently blocks somatic pain after abdominalwall surgery

. It providesadequate postoperative pain relief following various abdominal surgeries TAP block can reduce pain scores, opioid consumption, and the incidence of opioid-related complications after abdominal surgery.

The duration of the TAP block is limited to theeffect of the administered LAs. Various adjuvantmedications have been added to the LA to prolong theduration of TAP block and magnify its effects .

Perineural injection of steroids is reported to influence postoperative analgesia.

As a synthetic glucocorticoid, triamcinolone acetonide binds to and activates the glucocorticoid receptor to produce anti-inflammatory responses,such as down-regulating pro-inflammatory cytokine expression , preventing prostaglandin and leukotriene synthesis and release of arachidonic acid, and activating anti-inflammatory transcription factors such as lipocortins

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for major open abdominal surgery
* American Society Anesthesiologists (ASA) physical status I to II

Exclusion Criteria:

* Patient refusal.
* Morbidly obese patients.
* Patients with uncontrolled diabetes.
* Severe or uncontrolled renal, hepatic or endocrinal diseases.
* Pregnancy, post-partum or lactating females
* Allergy to one of the agents used.
* Recent (less than six months) use of glucocorticoids for at least two weeks

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
analgesic effect of Triamcinolone and Methylprednisolone In Ultrasound Guided Transversus Abdominis Plane Block ( Tap Block ). | 24 hours after surgery
  visual analogue scale for assessement of pain from 0 to 10 is used where 0 is no pain and 10 is maximum pain

SECONDARY OUTCOMES:
occurance of complication | 24 hours after surgery
  nausea vomiting hemodynamic changes

CONTACTS AND LOCATIONS:
Overall Officials: marwa M elegemazy, master, Principal Investigator — Mansoura University; ghada f amer, M.D, Study Director — associate professor of anesthesia; Eiad a ramzy, M.D, Study Chair — associate professor of anesthesia; abdelaziz a motaweaa, M.D, Study Chair — professor of anesthesia
Locations (1):
- Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No